CLINICAL TRIAL: NCT03965806
Title: Awareness About Field of Anaesthesiology and Role of Anaesthetist Among General Population of Ireland
Brief Title: Awareness About Anaesthesiology AND Role of Anaesthetist
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Our Lady of Lourdes Hospital, Drogheda (Other Government)
Responsible Party: Principal Investigator, SHANKAR LAL, SHANKAR, Our Lady of Lourdes Hospital, Drogheda
Other Study IDs: u2know1T
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: SURVEY
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SURVEY — SURVEY

SUMMARY:
INTRODUCTION:

Anaesthesia is a relatively new specialty as compared to medicine and surgery(1). Lack of public exposure and direct patient interaction have led to limited knowledge regarding anesthesiology among patients (2, 3). Status of anesthesiologist and anesthesiology in the eyes of public has always been a problem. Recent advancement in the field of anesthesiology has led to progress in surgical techniques and procedures, it is not always given its due share in media(2). Although professional bodies around the world are trying to improve awareness about anesthesiology, patient's knowledge about anesthesiology and anesthesiologist is largely inaccurate (4-6).

Studies done in developed countries have shown that patients have limited knowledge about role of anesthesiologist outside the operating room (2, 5, 7 ). A study done in India in 2009 shows that there was a wide spread ignorance about anesthesiology and role of anesthesiologist in general public(6). A survey done in Pakistan in 1999 showed that only 56% patients identified anesthesiologist as a doctor(4). Another study done in 2004 showed that 82% patients knew that anesthesiologist is a doctor but more than fifty percent had no idea about their other responsibilities in the hospital(8).

In recent past there may be an increase in awareness about anesthesiology because of explosive growth in media and internet (3). Whether this reflects on patient's knowledge needs to be determined. This information is important for establishing good patient doctor relationship and further efforts to educate general public about the importance of anesthesiology and role of anesthesiologist in health care.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to evaluate the current knowledge regarding field of anesthesiology and role of anesthesiologist in general population of Ireland.

Operational definitions:

Knowledge:

Knowledge of patients will be defined as the percentage of patients giving correct answers to a questionnaire consisting of questions modified from previous studies and other added questions (2-8). Patients giving 66% (8 out of 12) correct answers to the questionnaire will be considered to have knowledge of anesthesiology and anesthesiologist.

Methodology:

Study settings:

Study will be conducted among general population visiting or working in our lady of Lourdes Hospital.

Duration of study:

Study will be conducted over a period of two to three months after the approval of study.

Study design:

Cross-sectional study.

Sample size:

Sample size is calculated using WHO Sample Size Calculator. In a previously study(6) , knowledge regarding anesthesiologist and anesthesiology was about 51.52% therefore 384 patients will be include in this study to estimate knowledge within 5 percent point (margin of error) of the true value (51.52%) with 95% confidence interval.

Sampling technique:

Non-probability purposive sampling.

Inclusion criteria:

1. People visiting or working in our lady of Lourdes hospital.
2. Age 18 and above.
3. Both male and female

Exclusion criteria:

1. People refusing to give consent.
2. Pediatric patients (patients up to age of 16years).
3. Language barrier.
4. Patient unable to understand the questions due to disability.
5. Patients who are doctors.

Data collection:

After getting approval from the hospital .All subjects fulfilling the criteria will be enrolled in the study after taking informed consent. Patients will be interviewed by the preoperative SHO/Registrar or principal investigator in hospital. Each interview will last for 10-20min and will be based on attached questionnaire.

Questionnaire:

Questionnaire consist of questions modified from previous studies and added questions (2-9). It has two parts; demographics i.e. age, gender, educational level, occupation, previous anaesthesia experience and type of surgery, second part will consist of 12 questions about anesthesiology and anesthesiologist. Patients giving correct response to 8 out of 12 questions will be considered to have knowledge.

Data analysis:

All statistical analysis will be performed using statistical packages for social science version 19 (SPSS Inc., Chicago, IL). Frequency and percentage will be computed for gender, type of surgery, education level, previous surgery, Patient's knowledge about anesthesiology and anesthesiologist. Mean and standard deviation will estimated for age. Stratification will be done to control effect modifiers like gender, age, education level, previous surgery to observed Patient's knowledge about anesthesiology and anesthesiologist through chi-square test. p≤0.05 will be considered as significant.

References:

1. JM Klafta MR. Current understanding of patients' attitudes toward and preparation for anesthesia: a review. Anesthesia & Analgesia. 1996.
2. LM Calman AM, S Evron, T Ezri. Current understanding of the patient's attitude toward the anesthetist's role and practice in Israel: effect of the patient's experience. Journal of clinical anesthesia. 2003.
3. Seetharaman Hariharan MD LM-C, Deryk Chen. Patient perception of the role of anesthesiologists: a perspective from the Caribbean. Journal of Clinical Anesthesia 2006;18:504-9.
4. Khan F HS, Zaidi A. Patients view of the anaesthetist in a developing country. J Pak Med Assoc. 1999;49(1):4-7.
5. A. R. BRAUN KL, C. MORGAN, S. BUGLER. Patients' knowledge of the qualifications and roles of anaesthetists. Anaesth Intensive Care 2007;35 (4):570-4.
6. S K Mathur SKDaSJ. Knowledge about Anaesthesia and Anaesthesiologist Amongst General Population in India. Indian J Anaesth. 2009 April;53(2 ):179-86.
7. H. TOHMO HP, H. ILLMAN. The work, duties and prestige of Finnish anesthesiologists: patients' view. Acta Anaesthesiol Scand 2003;47:664-6.
8. Ahsan Ul Haq WA, Mubeen M. A survey of patients awareness about the peri-operative role of Anesthetists. Biomedica. 2004;20(1):5-9.
9. K Shevde GP. A survey of 800 patients' knowledge, attitudes, and concerns regarding anesthesia. Anesthesia & Analgesia. 1991;73.:190-8.

QUESTIONNAIRE AWARENESS ABOUT FIELD OF ANAESTHESIOLOGY AND ROLE OF ANAESTHETISTS AMONG GENERAL POPULATION OF IRELAND.

STUDY I.D:_______ VERBAL CONSENT TAKEN:

Age: __________________ years Gender: Male Female

Educational Level:

* Primary school education.
* Secondary school education.
* Intermediate.
* Graduate.
* Post graduate.

OCCUPATION:

* Health care professionals (other than doctors)
* Others (specify)_________________________ Previous Surgery: Yes No

KNOWLEDGE:

1. Have you heard about anaesthesia before: Yes No

   • If yes then where: TV Newspaper Internet Others______________
2. Has your surgeon told you anything about anaesthesia: Yes No
3. Are there different types of anaesthesia: Yes No

   • If yes what is the most common type of anaesthesia:

   General Spinal/epidural Local
4. Anesthesiology is a separate specialty: Yes No
5. How is patient kept asleep during surgery:

   Tablets I.V injections Gases Injection
6. Anaesthesia is provided by:

   Doctor Nurse Technician
7. How many years of training does anesthesiologist have 1 2 3 4 5 6
8. Perioperative well-being of patient is responsibility of:

   Surgeon Anesthesiologist Both
9. What does anesthesiologist do in operating room:

   Give drugs Monitors the patient Helps the surgeon Don't know Do paper work
10. Who ensures your well-being (BP, heart rate, ECG, respiration) in the operating room:

    Nurse Anesthesiologist Surgeon Technician
11. Who looks after the patient in recovery room:

    Nurse alone Nurse supervised by Anesthestist Nurse supervised by surgeon
12. In what areas in the hospital does the anesthesiologist take care of patients? Operating room (only) Intensive care unit (ICU) In pain management services and pain clinic In obstetric unit (labour epidural) In emergency department In medical research and education Don't Know

Number of correct answers: _________

Visit to preoperative anaesthesia clinic is important: Yes No Do you want further information about anaesthesia: Yes No Are you afraid of anaesthesia: Yes No

Who do you think is more important :

Surgeon Anesthesiologist Both are equal

ELIGIBILITY:
Inclusion Criteria:

1. People visiting or working in our lady of Lourdes hospital.
2. Age 18 and above.
3. Both male and female

Exclusion Criteria:

1. People refusing to give consent.
2. Pediatric patients (patients up to age of 16years).
3. Language barrier.
4. Patient unable to understand the questions due to disability.
5. Patients who are doctors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Population of Ireland visiting Hospital or Working in Our Lady of Lourdes Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
The objective of this study is to evaluate the current knowledge regarding field of anesthesiology and role of anesthesiologist in general population of Ireland. | 2 TO 3 MONTHS
  SURVEY

CONTACTS AND LOCATIONS:
Overall Officials: SHANKAR LAL, MBBS/FCPS, Principal Investigator — Our Lady of Lourdes Hospital
Locations (1):
- Our Lady of Lourdes Hospital, Drogheda, Louth, Ireland

IPD SHARING:
Plan to Share IPD: Undecided